CLINICAL TRIAL: NCT01924585
Title: Prospective Observational Study of Patients Aged >=60 Years Undergoing Major Gastrointestinal Surgery With 1 Year Follow-up
Brief Title: Surgery in Persons of Older Age
Acronym: SAGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 12/LO/1042-SAGE
Record Dates: First submitted 2013-08-12; First posted 2013-08-16 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2012-08

CONDITIONS: Colorectal Disorders; Surgery; Old Age; Debility; Quality of Life; Complications
Keywords: Colorectal; Surgery; Frailty; Elderly; Quality of Life
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Preoperative serum and urine sample.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Frail patient: Patients will be stratified into groups frail and non-frail based on pre-operative frailty and disability.

SUMMARY:
Surgery in persons of older AGE (SAGE) is an observational study of patients aged 60 years and older undergoing major colorectal surgery. That is to say we are looking at how older patients recovery following surgery, and that patients who volunteer to take part will absolutely not have any changes made to patients planned treatment or surgery.

Patients (identified by their Consultant) will be asked if they would like to participate in the study, agreeing to undertake an additional questionnaire, blood test, provide a urine specimen and several basic physical tests during the pre-assessment visit taking an additional 30-45 minutes.

This will not affect their treatment in any way. Participation is voluntary.

At the time of the pre-assessment process the patient will then be approached by a researcher, who will explain the study in more detail and obtain written consent.

The questionnaire is a combination of questions, which have been used in other similar studies and may be used to identify people who are fitter than others to undergo surgery. These questions are not too dissimilar to those that may be asked during the pre-assessment process. In fact some hospitals use some of these questions (but not usually all) routinely during a hospital admission process.

Several basic physical tests will be performed: hand grip strength test and some basic walking and chair rising tests. These will be supervised by the trained researcher to ensure they are carried out safely.

A small blood sample (20ml) will be obtained, ideally at the same time as blood is taken for the standard pre-operative assessment process. We will also take urine specimens. The blood sample and urine specimens will be saved for tests later. There are several potential blood and urine tests that may be related to physical frailty/impairment and the aging process.

The patient will undergo surgery as planned and be discharged from hospital. No researcher will interfere with the planned care or conduct any data collection at this point.

At approximately 1. 3, 6 and 12 months following surgery the patient will be asked to complete the questionnaire either in person, by phone or mail. If reviewed in a clinic at the time of their postoperative follow-up checks, then we will repeat the basic physical tests again also.

The patient's notes will be reviewed by a researcher (who is also a doctor) to see what operation was performed, the length of hospital stay, and if any problems developed. The patients GP may also be contacted if additional information is required.

This study, while based on several others, is the first of its kind to see how persons recover after surgery being assessed over one year.

We will recruit for 18 months across two hospitals aiming to recruit 200 patients during this time.

DETAILED DESCRIPTION:
Background

Lifespans are increasing and the proportion of elderly persons undergoing surgery is increasing[1]. As clinicians we need to accurately communicate the risks of major surgery to our patients. Traditional risk prediction tools such as Physiologic and operative Severity Score for the enumeration of Mortality and Morbidity (POSSUM) estimate short-term outcomes[2]. Patients have the right to know the likely outcomes beyond the 30-day perioperative period, including life expectancy, long-term complications, level of independence and quality of life[3].

Based on a systematic review of the literature we have previously reported on the paucity of studies evaluating longer-term outcomes in persons of advanced age undergoing major surgery[4].

Our group has previously reported, from analysis performed on an English administrative dataset, that patients face comparatively high mortality of 29% at one year following colorectal surgery when performed as an emergency[5]. Furthermore, we have published findings, again from national datasets, that patients 75-80 years of age undergoing colorectal resection in the elective setting also face substantial mortality of 16% at one-year, and over a third of patients aged >89 years who underwent surgery did not survive one-year[6].

Frailty, a distinct entity from co-morbidity, is recognized as an independent contributor to mortality in elderly surgical patients[7-10]. Thus we need to improve preoperative risk stratification for geriatric patients. Such systems may include frailty assessment and relevant predictive biomarkers. Thus we can then target additional healthcare resources towards the most frail and vulnerable elderly patients to mitigate against the risks of postoperative complications and death[11].

Preoperative optimisation strategies [12-14], careful intraoperative monitoring and postoperative care within the high dependency setting may reduce the frequency of postoperative complications, accelerate recovery and improve short-term outcomes. Furthermore, we need a collaborative research with elderly care and community physicians to determine whether ongoing postoperative community rehabilitation can offset the late risk of death associated with major surgery and further improve long-term survival.

Rationale for Current Study: Research Question

What preoperative parameters can be used to predict patient centered outcomes (survival, complications, functional independence, quality of life) in older persons undergoing major gastrointestinal elective surgery in the intermediate term?

Hypotheses

Traditional POSSUM scoring systems will not reliably predict outcomes at 1 year in elderly persons.

Patients determined to be frail preoperatively will have worse outcomes at 1 year, in terms of survival, postoperative complications, level of independence and quality of life.

Study Objectives

To identify the preoperative parameters that will predict 1 year outcomes in patients aged ≥60 years undergoing major gastrointestinal elective surgery.

Parameters include comprehensive geriatric assessment (i.e. a preoperative questionnaire of validated instruments assessing the dimensions of co-morbidities, activities of daily living, nutrition, cognitive function, emotional status, fatigue and performance status).

Furthermore patients will be asked to undergo a series of simple physical exercises (hand grip strength, timing up and go, 15 feet timing walking test, and 6 minute walking test).

Preoperative serum results will also be incorporated. Additional blood and urine samples will be obtained preoperative for later metabolic profiling.

Questionnaire, physical tests and biological sampling with be assessed at the time of the preoperative assessment process, or at another time preoperatively at the patients convenience.

Serum samples will be only obtained preoperatively. Urine samples may be collected following surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 60 years or older years undergoing elective major colorectal surgery.

Exclusion Criteria:

* Patients aged <60 years at time of operation.
* Severe cognitive impairment (Mini-mental score <18).
* Non-English language speaker.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 60 years or more, undergoing elective colorectal surgery (laparoscopic or open).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | Up to 1 Year Postoperatively
  Time to return to preoperative quality of life / level of functional independence.

SECONDARY OUTCOMES:
Complications | 30 days
  Clavien-Dindo complications
All Cause Mortality | 30 days postoperatively
Length of Hospital Stay | Average 5-10 days
Reoperation/reintervention | 30 day postoperatively
Re-admission | 30 days post-operatively
Discharge destination | 30 days post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Nigel M Bagnall, MBChB MRCS, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - St Mary's Hospital, London, London
  - St Mark's Hospital, Northwick Park NHS Trust, Harrow, Middlesex

REFERENCES:
- [Background] Etzioni DA, Liu JH, Maggard MA, Ko CY. The aging population and its impact on the surgery workforce. Ann Surg. 2003 Aug;238(2):170-7. doi: 10.1097/01.SLA.0000081085.98792.3d. PMID 12894008
- [Background] Al-Homoud S, Purkayastha S, Aziz O, Smith JJ, Thompson MD, Darzi AW, Stamatakis JD, Tekkis PP. Evaluating operative risk in colorectal cancer surgery: ASA and POSSUM-based predictive models. Surg Oncol. 2004 Aug-Nov;13(2-3):83-92. doi: 10.1016/j.suronc.2004.08.006. PMID 15572090
- [Background] Grocott MP, Pearse RM. Prognostic studies of perioperative risk: robust methodology is needed. Br J Anaesth. 2010 Sep;105(3):243-5. doi: 10.1093/bja/aeq207. No abstract available. PMID 20716567
- [Background] Mamidanna R, Almoudaris AM, Faiz O. Is 30-day mortality an appropriate measure of risk in elderly patients undergoing elective colorectal resection? Colorectal Dis. 2012 Oct;14(10):1175-82. doi: 10.1111/j.1463-1318.2011.02859.x. PMID 21999306
- [Background] Faiz O, Brown T, Bottle A, Burns EM, Darzi AW, Aylin P. Impact of hospital institutional volume on postoperative mortality after major emergency colorectal surgery in English National Health Service Trusts, 2001 to 2005. Dis Colon Rectum. 2010 Apr;53(4):393-401. doi: 10.1007/DCR.0b013e3181cc6fd2. PMID 20305437
- [Background] Faiz O, Haji A, Bottle A, Clark SK, Darzi AW, Aylin P. Elective colonic surgery for cancer in the elderly: an investigation into postoperative mortality in English NHS hospitals between 1996 and 2007. Colorectal Dis. 2011 Jul;13(7):779-85. doi: 10.1111/j.1463-1318.2010.02290.x. Epub 2010 Apr 19. PMID 20412094
- [Background] Makary MA, Segev DL, Pronovost PJ, Syin D, Bandeen-Roche K, Patel P, Takenaga R, Devgan L, Holzmueller CG, Tian J, Fried LP. Frailty as a predictor of surgical outcomes in older patients. J Am Coll Surg. 2010 Jun;210(6):901-8. doi: 10.1016/j.jamcollsurg.2010.01.028. Epub 2010 Apr 28. PMID 20510798
- [Background] Tan KY, Kawamura YJ, Tokomitsu A, Tang T. Assessment for frailty is useful for predicting morbidity in elderly patients undergoing colorectal cancer resection whose comorbidities are already optimized. Am J Surg. 2012 Aug;204(2):139-43. doi: 10.1016/j.amjsurg.2011.08.012. Epub 2011 Dec 16. PMID 22178483
- [Background] Sundermann S, Dademasch A, Rastan A, Praetorius J, Rodriguez H, Walther T, Mohr FW, Falk V. One-year follow-up of patients undergoing elective cardiac surgery assessed with the Comprehensive Assessment of Frailty test and its simplified form. Interact Cardiovasc Thorac Surg. 2011 Aug;13(2):119-23; discussion 123. doi: 10.1510/icvts.2010.251884. Epub 2011 Mar 4. PMID 21378017
- [Background] Robinson TN, Wu DS, Stiegmann GV, Moss M. Frailty predicts increased hospital and six-month healthcare cost following colorectal surgery in older adults. Am J Surg. 2011 Nov;202(5):511-4. doi: 10.1016/j.amjsurg.2011.06.017. Epub 2011 Sep 3. PMID 21890098
- [Background] Pearse RM, Holt PJ, Grocott MP. Managing perioperative risk in patients undergoing elective non-cardiac surgery. BMJ. 2011 Oct 5;343:d5759. doi: 10.1136/bmj.d5759. No abstract available. PMID 21976704
- [Background] Jack S, West M, Grocott MP. Perioperative exercise training in elderly subjects. Best Pract Res Clin Anaesthesiol. 2011 Sep;25(3):461-72. doi: 10.1016/j.bpa.2011.07.003. PMID 21925410
- [Background] Carli F, Charlebois P, Stein B, Feldman L, Zavorsky G, Kim DJ, Scott S, Mayo NE. Randomized clinical trial of prehabilitation in colorectal surgery. Br J Surg. 2010 Aug;97(8):1187-97. doi: 10.1002/bjs.7102. PMID 20602503
- [Background] Hennis PJ, Meale PM, Grocott MP. Cardiopulmonary exercise testing for the evaluation of perioperative risk in non-cardiopulmonary surgery. Postgrad Med J. 2011 Aug;87(1030):550-7. doi: 10.1136/pgmj.2010.107185. Epub 2011 Jun 21. PMID 21693573